CLINICAL TRIAL: NCT03364413
Title: Behavioral Assessment of the Brain Response to Bioactive Food Components Using Electroretinography (Brain's Response to Chocolate)
Brief Title: Brain's Response to Chocolate
Status: Completed | Type: Observational
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: Drexel University (Other)
Responsible Party: Sponsor
Other Study IDs: GFHNRC217
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Chocolate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chocolate: Participants will be asked to taste commercially available chocolate varying in sugar, fat and percent cocoa (milk, 70%, 85% and 90% cocoa).
  Interventions: Other: Chocolate

INTERVENTIONS:
Other: Chocolate — Participants will be asked to taste commercially available chocolate varying in sugar, fat and percent cocoa (milk, 70%, 85% and 90% cocoa).

SUMMARY:
The purpose of this study is to test how the brain responds when individuals eat enjoyable foods such as chocolate. Eating certain foods can make one want to keep eating even when feeling full, caused by dopamine in the brain. The researchers believe this dopamine response can be measured by looking at the individual's eye.

DETAILED DESCRIPTION:
With obesity at an all-time high, understanding eating behavior beyond physical need is a priority. Food reinforcement is driven by central dopamine activity. However, objective measurement of brain dopamine-related behavioral events is hindered by the lack of non-invasive, accessible techniques that are amenable to testing in a "naturalistic" environment. The goal of this project is to develop a non-invasive, accessible methodology to measure dopaminergic responses to food in a natural setting. This research will use a novel, hand-held electroretinograph (ERG) that does not require eye dilation and uses a skin electrode to measure retinal dopamine activity. Previous work establishes that retinal dopamine activity can be used as a proxy for central dopamine function. The ability to assess both subjective behavioral variables and central dopaminergic responses simultaneously will provide an ideal approach for innovative studies of the control of eating behavior.

ELIGIBILITY:
Inclusion Criteria:

* body mass index 20-30 kg/m2
* free of any major illness or disease

Exclusion Criteria:

* food allergies
* participation in a weight loss diet or exercise program
* pregnancy
* lactation
* metabolic illness or disease (diabetes, renal failure, thyroid illness, hypertension)
* eye illness or disease (narrow angle glaucoma, macular degeneration, retinal detachment, cataracts)
* psychiatric, neurological or eating disorders (schizophrenia, depression, Parkinson's Disease, Huntington's Disease, cerebral palsy, stroke, epilepsy, anorexia nervosa or bulimia nervosa)
* take prescription medications except for oral contraceptives or antihyperlipidemia agents

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Retinal dopamine response to oral stimuli | 30 minutes
  Electroretinograph beta wave amplitude will increase in response to increases in the amount of sugar in the chocolate
Psychoactive Effects Questionnaire in response to oral stimuli | 30 minutes
  The number of positive responses on the Psychoactive Effects Questionnaire will increase in response to increases in the sugar content of the chocolate

SECONDARY OUTCOMES:
Scores on the Binge Eating Scale will correlate with the retinal dopamine and Psychoactive Effect Questionnaire responses | 30 minutes
  Individual changes in the retinal dopamine response and the number of positive responses on the Psychoactive Effects Questionnaire will correlate with individual scores on the Binge Eating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Shanon Casperson, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Casperson SL, Lanza L, Albajri E, Nasser JA. Increasing Chocolate's Sugar Content Enhances Its Psychoactive Effects and Intake. Nutrients. 2019 Mar 12;11(3):596. doi: 10.3390/nu11030596. PMID 30870996